CLINICAL TRIAL: NCT01536977
Title: Early Behavioral Intervention in BMT Recipients With Sleep Disturbance: Assessing Its Impact on Quality of Life, Fatigue and Cognitive Function
Brief Title: Phase II Early Behavioral Intervention in BMT w/ Sleep Disturbance-Assess QOL+Fatigue+Cognitive f(x)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Oxana Palesh, Assistant Professor of Psychiatry and Behavioral Science, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BMT242; NCI-2012-00117 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SU-11112011-8650 (Other: Stanford University)
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Cognition Disorders; Fatigue; Sleep Disorders; Other Complications of Bone Marrow Transplant
Keywords: quality of life
MeSH Terms: conditions — Cognition Disorders; Fatigue; Sleep Wake Disorders | interventions — Mental Status and Dementia Tests; Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (BBT-I) (Experimental): Patients complete the BBT-I, comprising the following modules: 1) "What to expect" in terms of fatigue and insomnia as it occurs with cancer and cancer treatment; 2) A review of the Spielman Model of insomnia; 3) A discussion (based on the Spielman Model) regarding how insomnia and fatigue may co-occur and interact in the context of cancer and cancer treatment; 4) An introduction to the concept and practice of Stimulus Control Therapy; 5) An introduction to Sleep Scheduling Specifically modified for cancer patients; 6) Sleep Compression; and 7) Concomitant Medications and Substance Use.
  Interventions: Other: quality-of-life assessment; Other: questionnaire administration; Behavioral: management of therapy complications; Behavioral: cognitive assessment; Behavioral: educational intervention

INTERVENTIONS:
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies
Behavioral: management of therapy complications — Undergo BBT-I
  Other Names: complications of therapy, management of
Behavioral: cognitive assessment — Ancillary studies
Behavioral: educational intervention — Undergo BBT-I
  Other Names: intervention, educational

SUMMARY:
This pilot clinical trial studies early brief behavioral intervention in treating sleep disturbance and improving quality of life in patients undergoing bone marrow transplant (BMT). A brief behavioral intervention may reduce symptoms of insomnia and fatigue and improve quality of life and cognitive function in patients undergoing BMT

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To provide preliminary data on the feasibility and efficacy of brief behavioral treatment for insomnia (BBT-I) on insomnia in hematopoietic cell transplant (HCT) recipients.

SECONDARY OBJECTIVES:

I. To provide preliminary data on the influence of BBT-I on cancer-related fatigue (CRF) and cognitive status in BMT recipients.

II. To provide preliminary data on the influence of BBT-I on quality-of-life (QOL) in BMT recipients.

OUTLINE:

Patients complete the BBT-I, comprising the following modules: 1) "What to expect" in terms of fatigue and insomnia as it occurs with cancer and cancer treatment; 2) A review of the Spielman Model of insomnia; 3) A discussion (based on the Spielman Model) regarding how insomnia and fatigue may co-occur and interact in the context of cancer and cancer treatment; 4) An introduction to the concept and practice of Stimulus Control Therapy; 5) An introduction to Sleep Scheduling Specifically modified for cancer patients; 6) Sleep Compression; and 7) Concomitant Medications and Substance Use.

After completion of study treatment, patients are followed up at 1 month.

ELIGIBILITY:
Patients proceeding to BMT within the Stanford Adult BMT program will be screened for eligibility

Inclusion Criteria:

* Patient is scheduled to receive bone marrow transplantation.
* Patient has a diagnosis of Non-Hodgkin's Lymphoma
* Patient is at least 21 years old
* Patient is able to understand written and spoken English
* has preferred sleep phase between 9:00 pm and 3:00 am and a habitual rise time between 4:00 am and 11:00 am
* Patient receives a score of 8 or more on the Insomnia Severity Index or takes sleep medications 3 times a week

Exclusion criteria:

* Has an unstable medical or psychiatric illness (Axis I - current or within the last 5 years)
* Existing cognitive disability
* Is currently pregnant or nursing
* Has a history of substance abuse or meets criteria for current alcohol abuse or dependence
* Has a self-reported history of chronic pre-existing insomnia, sleep apnea or RSL syndrome

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Feasibility and efficacy of BBT-I on insomnia in HCT recipients as calculated by means, standard deviations and effect sizes on the Insomnia Severity Inventory (ISI) total score variable | Baseline
  The analysis will use longitudinal models with time as predictor and insomnia severity (ISI total score) as the dependent variable.
Feasibility and efficacy of BBT-I on insomnia in HCT recipients as calculated by means, standard deviations and effect sizes on the ISI variable | 6 weeks post-intervention
  The analysis will use longitudinal models with time as predictor and insomnia severity (ISI total score) as the dependent variable.

SECONDARY OUTCOMES:
Influence of BBT-I on CRF and cognitive status in BMT recipients | Baseline
Influence of BBT-I on CRF and cognitive status in BMT recipients | 6 weeks post-intervention
Influence of BBT-I on QOL in BMT recipients | Baseline
Influence of BBT-I on QOL in BMT recipients | 6 weeks post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Oxana Palesh, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States